CLINICAL TRIAL: NCT05815433
Title: Comparing Impacts of Donor Human Milk to Formula Supplementation on the Gut Microbiome of Full-term Infants Exposed to Antibiotics in Labour: A Pilot Randomized Controlled Trial
Brief Title: Comparing Impacts of Donor Human Milk to Formula Supplementation on the Gut Microbiome of Full-term Infants
Acronym: PPDHM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of British Columbia (Other); University of Victoria (Other); NorthernStar Mothers Milk Bank (Unknown)
Responsible Party: Principal Investigator, Meredith Brockway, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMS23-99633743
Record Dates: First submitted 2023-03-15; First posted 2023-04-18 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Microbial Colonization
Keywords: Sleep; Microbiome; Growth; Postpartum depression; Maternal anger; Breastfeeding; Self-efficacy
MeSH Terms: conditions — Communicable Diseases; Depression, Postpartum; Breast Feeding

STUDY DESIGN:
Intervention Model Description: An experimental study design in which each participants will be randomized to one of two groups (intervention [DHM] or standard care/control [formula])
Who Masked: Outcomes Assessor
Masking Description: Assessors who are conducting the microbial analysis and statistical analysis will not be aware of which group is intervention and which is control. These groups will be assigned a number (Group 1; Group 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donor Human Milk (Experimental): Infants randomized to the intervention group will receive DHM each time supplementation is required for the first 7 days of life.
  Interventions: Other: Donor Human Milk - Nutritional Replacement
- Standard Care (Infant Formula) (No Intervention): Infants randomized to the standard care group will receive formula each time supplementation is required for the first 7 days of life.

INTERVENTIONS:
Other: Donor Human Milk - Nutritional Replacement — All DHM in North America is pasteurized and provided through certified milk banks regulated by the Human Milk Banking Association of North America. DHM for this study will be obtained from the NorthernStar Mothers Milk Bank (NMMB). The milk is pasteurized and rigorously tested according to Human Milk Banking of North America guidelines. In Canada, DHM is categorized as food or nutritional therapy and the milk bank is monitored and certified by the Canadian Food Inspection Agency. The product used for this study will be the same product that is provided to other hospital units (mainly the neonatal intensive care units) in Alberta and around Canada. The product will not be modified or tampered with in any way.
  Arms: Donor Human Milk

SUMMARY:
The goal of this pilot randomized controlled trial (RCT) is to examine donor human milk (DHM) as a clinical intervention targeted at achieving beneficial microbiome signatures in full-term infants who are exposed to intrapartum antibiotic prophylaxis (IAP) therapy during labour. Secondarily, this study aims to compare the infant health outcomes of sleep and growth between groups to assess if these outcomes are mediated by infant feeding type or potential differences in microbial signatures. Finally, this study will compare maternal outcomes of depression, anger, breastfeeding self-efficacy and breastfeeding rates between groups.

The hypothesis of this study is: that replacing formula with DHM supplementation will minimize gut microbiome dysbiosis and foster homeostasis following supplementation. In addition, it is hypothesized that improved homeostasis will promote improved sleep and growth outcomes in participant infants. Finally, mothers whose infants receive DHM will have lower depression and anger scores and high breastfeeding self-efficacy and exclusive breastfeeding rates compared to mothers whose infants receive formula.

DETAILED DESCRIPTION:
Investigators propose to conduct a pilot clinical RCT in the postpartum hospital setting examining DHM as an intervention provided to full-term infants who are exposed to Group B Streptococcus (GBS) antibiotic prophylaxis during labour. Randomization of participant infants is currently an ethical practice because DHM supplementation is not standard practice in this population; infants receive formula if supplementation of mother's own milk (MOM) is required. Additionally, randomization will allow investigators to determine causal relationships between DHM supplementation compared to formula supplementation on the infant gut microbiome. Finally, conducting research in the clinical setting will allow for pragmatic assessment of DHM as an intervention, enhancing external validity and increasing the likelihood of its implementation into healthcare systems to improve healthcare quality.

Population: The population of interest is vaginally born, full-term infants who are exposed to antibiotics in labour through IAP and whose mothers are planning on breastfeeding.

Recruitment: Mothers greater than 37 weeks' gestation admitted to the postpartum unit who test positive for GBS and deliver vaginally will be screened for participation in the study by nurses on the postpartum unit. Approximately 20% of all pregnant mothers will test positive for GBS and Alberta Health Services protocol indicates that GBS-positive mothers are given intravenous antibiotics during labour. Only mothers who receive the complete Alberta Health Services protocol will qualify for the study. Upon recruitment and completion of informed consent, infants requiring supplementation of MOM will be randomized to the control or intervention group. Investigators will randomize 60 mother-infant dyads, providing adequate power to detect overall microbiome differences (~30 in each group).

Intervention - Donor Human Milk (DHM): Infants randomized to the intervention group will receive DHM each time supplementation is required for the first 7 days of life. The exposure time of 7 days was selected due to feasibility of DHM cost, and this is the period when breastfeeding is being established and most formula supplementation occurs. Infants in the control group will receive formula when supplementation is required (standard care). All DHM in North America is pasteurized and provided through certified milk banks regulated by the Human Milk Banking Association of North America and DHM for this study will be obtained from the NorthernStar Mothers Milk Bank (NMMB).

Data Collection, Analysis, and Outcomes: The primary outcome for this pilot study will result from comparisons of DHM to formula supplementation groups for differences in microbiome signatures, such as diversity, proportions of Bifidobacteria, and proportions of pathogenic organisms. Infant stool samples will be collected from soiled diapers at one, six and 12 weeks postpartum.

Secondary outcomes include infant growth, sleep, and breastfeeding outcomes that will be collected at one, six and 12 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Gestation greater than 37 weeks (full-term)
* Completion of antibiotic protocol for GBS during labour
* Vaginal delivery
* Intending on breastfeeding
* Consent for infant to receive DHM
* Working understanding (proficient in reading and understanding) English
* Mother has provided signed and dated informed consent and authorization to use protected health information, as required by national and local regulations.
* In the investigator's opinion, the subject mother understands and can comply with protocol requirements, instructions, and protocol-stated restrictions, and is likely to complete the study as planned.

Exclusion Criteria:

* Diagnosed with clinically significant major congenital malformation that will interfere with breastfeeding or growth
* No intention to breastfeed
* Receiving extended courses of antibiotics (beyond that of the IAP in labour)

Min Age: 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Infant gut microbiome - shallow shotgun metagenomics (RA) | one week postpartum
  Relative abundance
Infant gut microbiome - shallow shotgun metagenomics (RA) | six weeks postpartum
  Relative abundance
Infant gut microbiome - shallow shotgun metagenomics (RA) | twelve weeks postpartum
  Relative abundance
Infant gut microbiome - shallow shotgun metagenomics (alpha diversity) | one week postpartum
  alpha diversity of microbiome
Infant gut microbiome - shallow shotgun metagenomics (alpha diversity) | six weeks postpartum
  alpha diversity of microbiome
Infant gut microbiome - shallow shotgun metagenomics (alpha diversity) | twelve weeks postpartum
  alpha diversity of microbiome
Infant gut microbiome - shallow shotgun metagenomics (beta diversity) | one week postpartum
  beta diversity of microbiome
Infant gut microbiome - shallow shotgun metagenomics (beta diversity) | six weeks postpartum
  beta diversity of microbiome
Infant gut microbiome - shallow shotgun metagenomics (beta diversity) | twelve weeks postpartum
  beta diversity of microbiome

SECONDARY OUTCOMES:
Infant Sleep | Six weeks postpartum
  Brief Infant Sleep Questionnaire - Revised Short Form - Scores on each subscale and the total score are scaled from 0 to 100, with higher scores denoting better sleep quality, more positive perception of infant sleep, and parent behaviors that promote healthy and independent sleep.
Infant Sleep | Twelve weeks postpartum
  Brief Infant Sleep Questionnaire- Scores on each subscale and the total score are scaled from 0 to 100, with higher scores denoting better sleep quality, more positive perception of infant sleep, and parent behaviors that promote healthy and independent sleep.
Infant Growth - weight | one week postpartum
  Weight - in grams; weight and height will be combined to report BMI in kg/m^2
Infant Growth - length | one week postpartum
  Length - in centimeters; weight and height will be combined to report BMI in kg/m^2
Infant Growth - BMI | one week postpartum
  Body mass index - weight and height will be combined to report BMI in kg/m^2
Infant Growth - BMI | six weeks postpartum
  Body mass index - weight and height will be combined to report BMI in kg/m^2
Infant Growth - BMI | twelve weeks postpartum
  Body mass index - weight and height will be combined to report BMI in kg/m^2
Infant Growth - head | one week postpartum
  Head circumference - in centimeters
Infant Growth - weight | six weeks postpartum
  Weight- in grams; weight and height will be combined to report BMI in kg/m^2
Infant Growth- length | six weeks postpartum
  Length - in centimeters; weight and height will be combined to report BMI in kg/m^2
Infant Growth - head | six weeks postpartum
  Head circumference - in centimeters
Infant Growth - weight | Twelve weeks postpartum
  Weight- in grams; weight and height will be combined to report BMI in kg/m^2
Infant Growth- length | Twelve weeks postpartum
  Length - in centimeters; weight and height will be combined to report BMI in kg/m^2
Infant Growth - head | Twelve weeks postpartum
  Head circumference - in centimeters
Infant feeding | one week postpartum
  breastfeeding exclusivity - measured by 7-day infant feeding journal. Number of participants whose consume only breastmilk.
Infant feeding | six weeks postpartum
  breastfeeding exclusivity - measured by 7-day maternal recall. Number of participants whose consume only breastmilk.
Infant feeding | twelve weeks postpartum
  breastfeeding exclusivity- measured by 7-day maternal recall. Number of participants whose consume only breastmilk.
Maternal Depression | one week postpartum
  Edinburgh Postnatal Depression Screen - Range in score from 0 to 30; higher scores indicate worse outcomes
Maternal Depression | six weeks postpartum
  Edinburgh Postnatal Depression Screen - Range in score from 0 to 30; higher scores indicate worse outcomes
Maternal Depression | twelve weeks postpartum
  Edinburgh Postnatal Depression Screen -- Range in score from 0 to 30; higher scores indicate worse outcomes
Maternal Anger | one week postpartum
  LEVEL 2-Anger-Adult (PROMIS Emotional Distress-Anger- Short Form): Range in score from 5 to 25 with higher scores indicating greater severity of anger.
Maternal Anger | six weeks postpartum
  LEVEL 2-Anger-Adult (PROMIS Emotional Distress-Anger- Short Form): Range in score from 5 to 25 with higher scores indicating greater severity of anger.
Maternal Anger | twelve weeks postpartum
  LEVEL 2-Anger-Adult (PROMIS Emotional Distress-Anger- Short Form): Range in score from 5 to 25 with higher scores indicating greater severity of anger.
Maternal Breastfeeding Self-efficacy | one week postpartum
  Breastfeeding self-efficacy scale - short form: Total scores range from 14 to 70, with higher scores reflecting more significant levels of breastfeeding self-efficacy.
Maternal Breastfeeding Self-efficacy | six weeks postpartum
  Breastfeeding self-efficacy scale - short form: Total scores range from 14 to 70, with higher scores reflecting more significant levels of breastfeeding self-efficacy.
Maternal Breastfeeding Self-efficacy | twelve weeks postpartum
  Breastfeeding self-efficacy scale - short form: Total scores range from 14 to 70, with higher scores reflecting more significant levels of breastfeeding self-efficacy.
Maternal Anxiety | Baseline - (birth/enrolment)
  State - trait Anxiety inventory: Total scores range from 20 to 80 (each for state and trait), with higher scores indicating worse outcomes (higher anxiety).
Maternal Anxiety | six weeks postpartum
  State Anxiety inventory: Total scores range from 20 to 80, with higher scores indicating worse outcomes (higher anxiety).
Maternal Anxiety | twelve weeks postpartum
  State Anxiety inventory: Total scores range from 20 to 80, with higher scores indicating worse outcomes (higher anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Brockway, PhD RN, Principal Investigator — University of Calgary
Locations (1):
- Rockyview General Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon request

REFERENCES:
- [Background] Matenchuk BA, Mandhane PJ, Kozyrskyj AL. Sleep, circadian rhythm, and gut microbiota. Sleep Med Rev. 2020 Oct;53:101340. doi: 10.1016/j.smrv.2020.101340. Epub 2020 May 13. PMID 32668369
- [Background] Robertson RC, Manges AR, Finlay BB, Prendergast AJ. The Human Microbiome and Child Growth - First 1000 Days and Beyond. Trends Microbiol. 2019 Feb;27(2):131-147. doi: 10.1016/j.tim.2018.09.008. Epub 2018 Oct 24. PMID 30529020
- [Background] Tamburini S, Shen N, Wu HC, Clemente JC. The microbiome in early life: implications for health outcomes. Nat Med. 2016 Jul 7;22(7):713-22. doi: 10.1038/nm.4142. PMID 27387886
- [Background] Arrieta MC, Stiemsma LT, Amenyogbe N, Brown EM, Finlay B. The intestinal microbiome in early life: health and disease. Front Immunol. 2014 Sep 5;5:427. doi: 10.3389/fimmu.2014.00427. eCollection 2014. PMID 25250028
- [Background] Korpela K, de Vos WM. Infant gut microbiota restoration: state of the art. Gut Microbes. 2022 Jan-Dec;14(1):2118811. doi: 10.1080/19490976.2022.2118811. PMID 36093611
- [Background] Persaud RR, Azad MB, Chari RS, Sears MR, Becker AB, Kozyrskyj AL; CHILD Study Investigators. Perinatal antibiotic exposure of neonates in Canada and associated risk factors: a population-based study. J Matern Fetal Neonatal Med. 2015 Jul;28(10):1190-5. doi: 10.3109/14767058.2014.947578. Epub 2014 Aug 14. PMID 25053193
- [Background] Zimmermann P, Curtis N. Effect of intrapartum antibiotics on the intestinal microbiota of infants: a systematic review. Arch Dis Child Fetal Neonatal Ed. 2020 Mar;105(2):201-208. doi: 10.1136/archdischild-2018-316659. Epub 2019 Jul 11. PMID 31296695
- [Background] Stuivenberg GA, Burton JP, Bron PA, Reid G. Why Are Bifidobacteria Important for Infants? Microorganisms. 2022 Jan 25;10(2):278. doi: 10.3390/microorganisms10020278. PMID 35208736
- [Background] Liu Y, Qin S, Song Y, Feng Y, Lv N, Xue Y, Liu F, Wang S, Zhu B, Ma J, Yang H. The Perturbation of Infant Gut Microbiota Caused by Cesarean Delivery Is Partially Restored by Exclusive Breastfeeding. Front Microbiol. 2019 Mar 26;10:598. doi: 10.3389/fmicb.2019.00598. eCollection 2019. PMID 30972048
- [Background] Korpela K, Salonen A, Virta LJ, Kekkonen RA, de Vos WM. Association of Early-Life Antibiotic Use and Protective Effects of Breastfeeding: Role of the Intestinal Microbiota. JAMA Pediatr. 2016 Aug 1;170(8):750-7. doi: 10.1001/jamapediatrics.2016.0585. PMID 27294842
- [Background] Dai DLY, Petersen C, Hoskinson C, Del Bel KL, Becker AB, Moraes TJ, Mandhane PJ, Finlay BB, Simons E, Kozyrskyj AL, Patrick DM, Subbarao P, Bode L, Azad MB, Turvey SE. Breastfeeding enrichment of B. longum subsp. infantis mitigates the effect of antibiotics on the microbiota and childhood asthma risk. Med. 2023 Feb 10;4(2):92-112.e5. doi: 10.1016/j.medj.2022.12.002. Epub 2023 Jan 4. PMID 36603585
- [Background] Forbes JD, Azad MB, Vehling L, Tun HM, Konya TB, Guttman DS, Field CJ, Lefebvre D, Sears MR, Becker AB, Mandhane PJ, Turvey SE, Moraes TJ, Subbarao P, Scott JA, Kozyrskyj AL; Canadian Healthy Infant Longitudinal Development (CHILD) Study Investigators. Association of Exposure to Formula in the Hospital and Subsequent Infant Feeding Practices With Gut Microbiota and Risk of Overweight in the First Year of Life. JAMA Pediatr. 2018 Jul 2;172(7):e181161. doi: 10.1001/jamapediatrics.2018.1161. Epub 2018 Jul 2. Erratum In: JAMA Pediatr. 2018 Jul 1;172(7):704. doi: 10.1001/jamapediatrics.2018.2205. PMID 29868719
- [Background] Francis J, Mildon A, Stewart S, Underhill B, Ismail S, Di Ruggiero E, Tarasuk V, Sellen DW, O'Connor DL. Breastfeeding rates are high in a prenatal community support program targeting vulnerable women and offering enhanced postnatal lactation support: a prospective cohort study. Int J Equity Health. 2021 Mar 3;20(1):71. doi: 10.1186/s12939-021-01386-6. PMID 33658034
- [Background] Ho NT, Li F, Lee-Sarwar KA, Tun HM, Brown BP, Pannaraj PS, Bender JM, Azad MB, Thompson AL, Weiss ST, Azcarate-Peril MA, Litonjua AA, Kozyrskyj AL, Jaspan HB, Aldrovandi GM, Kuhn L. Meta-analysis of effects of exclusive breastfeeding on infant gut microbiota across populations. Nat Commun. 2018 Oct 9;9(1):4169. doi: 10.1038/s41467-018-06473-x. PMID 30301893
- [Background] Chong HY, Tan LT, Law JW, Hong KW, Ratnasingam V, Ab Mutalib NS, Lee LH, Letchumanan V. Exploring the Potential of Human Milk and Formula Milk on Infants' Gut and Health. Nutrients. 2022 Aug 29;14(17):3554. doi: 10.3390/nu14173554. PMID 36079814
- [Background] Peila C, Moro GE, Bertino E, Cavallarin L, Giribaldi M, Giuliani F, Cresi F, Coscia A. The Effect of Holder Pasteurization on Nutrients and Biologically-Active Components in Donor Human Milk: A Review. Nutrients. 2016 Aug 2;8(8):477. doi: 10.3390/nu8080477. PMID 27490567
- [Background] Merjaneh N, Williams P, Inman S, Schumacher M, Ciurte A, Smotherman C, Alissa R, Hudak M. The impact on the exclusive breastfeeding rate at 6 months of life of introducing supplementary donor milk into the level 1 newborn nursery. J Perinatol. 2020 Jul;40(7):1109-1114. doi: 10.1038/s41372-020-0657-6. Epub 2020 Mar 30. PMID 32231257
- [Background] Whipps MDM, Yoshikawa H, Demirci JR, Hill J. Estimating the Impact of In-Hospital Infant Formula Supplementation on Breastfeeding Success. Breastfeed Med. 2021 Jul;16(7):530-538. doi: 10.1089/bfm.2020.0194. Epub 2021 Jun 10. PMID 34115545
- [Background] Wiggins JB, Trotman R, Perks PH, Swanson JR. Enteral Nutrition: The Intricacies of Human Milk from the Immune System to the Microbiome. Clin Perinatol. 2022 Jun;49(2):427-445. doi: 10.1016/j.clp.2022.02.009. PMID 35659095
- [Background] McCune S, Perrin MT. Donor Human Milk Use in Populations Other than the Preterm Infant: A Systematic Scoping Review. Breastfeed Med. 2021 Jan;16(1):8-20. doi: 10.1089/bfm.2020.0286. Epub 2020 Nov 25. PMID 33237802
- [Background] Rao S, Esvaran M, Chen L, Keil AD, Gollow I, Simmer K, Wemheuer B, Conway P, Patole S. Probiotic supplementation in neonates with congenital gastrointestinal surgical conditions: a pilot randomised controlled trial. Pediatr Res. 2022 Oct;92(4):1122-1131. doi: 10.1038/s41390-021-01884-x. Epub 2022 Jan 3. PMID 34980887